CLINICAL TRIAL: NCT06874387
Title: Towards a Better Understanding of the Combination of Intermittent Hypoxia and Physical Exercise: Comparison of Effects on Cognitive and Cerebral Capacities in Middle-Aged Adults
Brief Title: Investigating the Combined Effects of Intermittent Hypoxia and Exercise on Cognitive and Cerebral Function in Middle-Aged Adults
Acronym: HYPOX-AGE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ayoub Boulares (Other)
Collaborators: University of Poitiers (Other); Laboratory MOVE, Faculty of Sport Sciences, University of Poitiers, France (Unknown)
Responsible Party: Sponsor-Investigator, Ayoub Boulares, Principal Investigator, PhD student, University of Poitiers
Organization: University of Poitiers (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HYPOX-AGE-2024-A00894-43
Record Dates: First submitted 2025-02-25; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Ability, General; Brain Health; Cerebral Oxygenation
Keywords: intermittent Hypoxia Training; Hypoxic Conditioning; Physical Activity; Exercise Intervention; Cognitive Function; Brain Health; Non-Pharmacological Interventions; Middle-Aged Adults; Healthy Aging; Cognitive Decline Prevention; Neuroplasticity
MeSH Terms: conditions — Motor Activity | interventions — Exercise; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-group trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Intermittent Hypoxia Only (Experimental): Participants in this arm will undergo a protocol of repeated cycles of hypoxia and normoxia. Each session will consist of alternating 5-minute hypoxic exposures with 5-minute normoxic intervals, for a total of approximately 30 minutes per session. Sessions will be held three times per week for six weeks (18 total sessions), and will be conducted at rest inside a hypoxic chamber under clinical supervision.
  Interventions: Other: Hypoxia, intermittent
- Physical exercise only (Experimental): Participants allocated to this arm will engage in a moderate-intensity aerobic exercise program (~60-70% of age-predicted maximum heart rate and based on a standardized scale of perceived exertion) three times per week for six weeks (total of 18 sessions). Each session will last approximately 30 minutes and may involve activities such as treadmill walking, cycling, or other forms of continuous aerobic exercise. The exercise intensity is monitored (e.g., via heart rate or perceived exertion) to ensure a moderate level of effort that is both safe and beneficial for overall cardiovascular and cognitive health.
  Interventions: Other: physical exercise
- Sequential Combination of Intermittent Hypoxia (IH) and Physical Activity (PA) (Experimental): Participants in this arm will undergo both Intermittent Hypoxia Training (IH) and Physical Activity (PA) within the same session, but in a sequential manner. The order of interventions (IH first or PA first) will be randomized to account for potential order effects. Each session consists of 30 minutes of IHT (5-minute hypoxia cycles, followed by 5-minute normoxic intervals, with SpO₂ maintained between 80% and 90%) and 30 minutes of moderate-intensity aerobic exercise (e.g., treadmill walking, cycling). Sessions will be held three times per week for six weeks (18 total sessions) and will be conducted under clinical supervision in a controlled environment.
  Interventions: Other: Hypoxia, intermittent; Other: physical exercise
- Simultaneous Combination of Intermittent Hypoxia (IH) and Physical Activity (PA) (Experimental): Participants in this arm will undergo Intermittent Hypoxia (IH) and Physical Activity (PA) simultaneously within the same session. During each session, participants will engage in moderate-intensity aerobic exercise (e.g., treadmill walking or cycling) while being exposed to IH. The total session duration will be 30 minutes, consisting of repeated cycles of 5 minutes of hypoxia followed by 5 minutes of normoxia, with SpO₂ maintained between 80% and 90% during hypoxic intervals. Sessions will be conducted three times per week for six weeks (18 total sessions) under clinical supervision in a controlled environment.
  Interventions: Other: Hypoxia, intermittent; Other: physical exercise
- Sham (Placebo) Intermittent Hypoxia (Placebo Comparator): Participants in this arm will undergo a sham (placebo) version of Intermittent Hypoxia (IH), where they will be exposed to normoxic air (FiO₂ ~20.9%) instead of actual hypoxia. The session structure will mimic the IH protocol, alternating between 5-minute "hypoxia" periods and 5-minute normoxia periods for a total of 30 minutes per session, but without a real reduction in oxygen levels. Sessions will be held three times per week for six weeks (18 total sessions) and will be conducted at rest inside a hypoxic chamber under clinical supervision.
  Interventions: Other: Sham (No Treatment) hypoxia

INTERVENTIONS:
Other: Hypoxia, intermittent — Moderate-Intensity Aerobic Exercise (~60-70% of maximum heart rate) and Intermittent Hypoxia (maintained between 80-90% during hypoxic phases)
  Other Names: hypoxic expousre
  Arms: Intermittent Hypoxia Only; Sequential Combination of Intermittent Hypoxia (IH) and Physical Activity (PA); Simultaneous Combination of Intermittent Hypoxia (IH) and Physical Activity (PA)
Other: physical exercise — Moderate-Intensity Aerobic Exercise (~60-70% of maximum heart rate)
  Arms: Physical exercise only; Sequential Combination of Intermittent Hypoxia (IH) and Physical Activity (PA); Simultaneous Combination of Intermittent Hypoxia (IH) and Physical Activity (PA)
Other: Sham (No Treatment) hypoxia — Exposure to normoxic air (FiO₂ ~20.9%) instead of actual hypoxia.
  Arms: Sham (Placebo) Intermittent Hypoxia

SUMMARY:
This study investigates whether intermittent hypoxia (IH) and physical activity (PA), either alone or in combination (simultaneously or sequentially), can improve cognitive function and brain health in middle-aged adults (50-65 years old). The hypothesis is that (1) each intervention alone (IHT or PA) provides cognitive benefits and (2) combining IHT with PA may yield additive or synergistic effects, particularly when administered simultaneously rather than sequentially. By comparing these distinct interventions, the study aims to determine which approach best preserves or enhances cognitive performance in middle-aged adults. Findings from this research may inform non-pharmacological strategies to promote healthy aging and reduce the risk of age-related cognitive decline.

DETAILED DESCRIPTION:
Rapid demographic aging worldwide is driving a surge in age-related conditions, including neurodegenerative diseases and cognitive disorders. Projections estimate that the number of people living with dementia could reach 78 million by 2030 and 139 million by 2050, underscoring the urgent need for effective, non-pharmacological strategies to preserve brain health. Intermittent hypoxia (IH) and physical activity (PA) are two promising interventions that may help prevent or mitigate cognitive decline. IH-an approach involving repeated cycles of reduced oxygen (11-16% FiO₂) followed by normoxic recovery-has shown benefits across diverse health domains (cardiovascular, metabolic, respiratory, and neurological), potentially through mechanisms such as the activation of Hypoxia-Inducible Factor (HIF), enhanced vascular endothelial growth factor (VEGF) production, and anti-apoptotic pathways. PA is widely recognized for its positive impact on overall health, including cognitive function and neuroplasticity.

The primary objective of this study is to evaluate the effects of IH and PA-administered individually, sequentially, or simultaneously-on cognitive performance and brain health in adults aged 50 to 65. The study will determine whether combining these interventions produces additive or synergistic benefits beyond those observed with each intervention alone. A total of approximately 176 participants will be enrolled and randomly assigned to one of five groups: (1) PA only, (2) IH only, (3) PA + IH sequentially, (4) PA + IH simultaneously, or (5) a control group receiving "placebo" hypoxia. Each participant will complete 18 sessions over a 6-week period (3 sessions per week), with sessions conducted in a hypoxic chamber at CIC 1402 and at the exercise testing facility of the University of Poitiers.

Outcome measures include comprehensive cognitive testing (global cognition, reaction time, executive function, and divided attention), assessments of autonomy (e.g., activities of daily living), and physiological parameters (e.g., SpO₂, cerebral oxygenation, heart rate, and blood pressure). Biomarker analysis will include brain-derived neurotrophic factor (BDNF), VEGF, irisin, and markers of HIF activation to elucidate the mechanisms underlying any observed improvements. Vascular function will be assessed using Doppler ultrasound and near-infrared spectroscopy (NIRS), and daily activity levels will be monitored with accelerometers.

Inclusion criteria require participants to be 50-65 years old, with a Montreal Cognitive Assessment (MoCA) score ≥24, no participation in other exercise interventions in the past 6 months, and no altitude exposure above 1,500 m in the preceding 3 months. Additional eligibility requirements include the absence of chronic kidney, cardiovascular, metabolic, neurological, or orthopedic disease, as well as no significant respiratory history. Exclusion criteria include active smoking, major cardiovascular complications within the last 3 months, severe hypertension, chronic respiratory insufficiency, diabetes, or any other condition that could compromise safety or study compliance. A qualified medical doctor will confirm eligibility during the inclusion process.

By evaluating different delivery methods of IH and PA, this research aims to identify the most effective, non-pharmacological approach to preserving-or potentially enhancing-cognitive function in middle-aged adults. Findings may contribute to targeted preventive strategies and novel therapeutic interventions, addressing the growing public health burden of age-related cognitive decline.

ELIGIBILITY:
* Inclusion Criteria:

  * Adults aged 50 to 65 years (male and female)
  * Montreal Cognitive Assessment (MoCA) score ≥ 24
  * No participation in any structured exercise intervention in the last 6 months
  * No exposure to altitudes above 1,500 m in the preceding 3 months
  * No chronic kidney, cardiovascular, metabolic, neurological, or orthopedic -disease
  * No history of significant respiratory conditions (e.g., asthma, exercise-induced -bronchospasm, dyspnea on exertion)
  * No current immunosuppressive treatment (e.g., corticosteroids, antidepressants)
  * No history of cancer or arthritis treatments
  * No recent blood donation (within the last 2 months)
  * Must be covered by a Social Security system or equivalent
  * Signed informed consent after receiving clear and transparent study information
  * Eligibility confirmed by a medical doctor during the inclusion process
* Exclusion Criteria:

  * Active smoking
  * Major cardiovascular complications within the last 3 months (e.g., myocardial i-infarction, unstable angina, severe arrhythmias)
  * Severe hypertension (≥180 mmHg systolic or ≥110 mmHg diastolic)
  * Chronic respiratory insufficiency (e.g., COPD, sleep apnea)
  * Diabetes mellitus
  * Need for continuous or intermittent oxygen therapy
  * Participation in another clinical study at the same time
  * Use of corticosteroids or other systemic immunosuppressants
  * Any condition compromising safety or study compliance, as determined by the medical team
  * Pregnancy or breastfeeding
  * Legal or administrative protections (e.g., individuals under guardianship, persons deprived of liberty)
  * High baseline physical activity levels (PASE score >90 indicating moderate-to-intense physical activity)

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — males and females
Enrollment: 176 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function: Montreal Cognitive Assessment (MoCA) | Baseline (Week 0),Week 1 (after 3 sessions), Week 6 (post-intervention, after session 18)
  1-Montreal Cognitive Assessment (MoCA)
  * Score Range: 0 to 30
  * Interpretation: Higher scores indicate better cognitive function.
Cerebral Oxygenation - Tissue Saturation Index (TSI) | Baseline (Week 0), Week 1 (after 3 sessions), Week 6 (post-intervention, after session 18)
  * Method: Near-Infrared Spectroscopy (NIRS)
  * Measure: Tissue Saturation Index (TSI), expressed as a percentage (%)
  * Interpretation: Higher TSI values indicate better cerebral oxygenation, reflecting efficient oxygen delivery and utilization in brain tissue.
Biomarker Analysis- Brain-Derived Neurotrophic Factor (BDNF) Levels | Baseline (Week 0), Week 1 (after 3 sessions), Week 6 (post-intervention, after session 18)
  * Method: Enzyme-Linked Immunosorbent Assay (ELISA)
  * Unit of Measure: pg/mL
  * Interpretation: Higher BDNF levels indicate greater neuroplasticity, neuronal survival, and cognitive function support.
Cerebral blood flow | Baseline (Week 0), Week 1 (after 3 sessions), Week 6 (post-intervention, after session 18)
  Method: Transcranial Doppler (TCD) Measures: Mean, systolic, and diastolic blood flow velocities in cerebral arteries.
  Interpretation: Higher flow velocities indicate increased cerebral perfusion, while reduced velocities may reflect impaired blood flow regulation or vascular resistance.
Cognitive Function: Stroop Test | Baseline (Week 0), Week 1 (after 3 sessions), Week 6 (post-intervention, after session 18)
  The Stroop Test is a widely used cognitive assessment tool designed to measure executive function, specifically selective attention, cognitive flexibility, and inhibitory control. It evaluates the ability to suppress automatic responses and manage conflicting information.
  -Score Range: Reaction Time (measured in milliseconds, ms): Represents the time taken to respond in each condition.
  Accuracy Percentage (%): Indicates the proportion of correct responses relative to total trials.
  -Interpretation: Lower reaction times indicate faster cognitive processing and improved efficiency in managing conflicting information.
  Higher accuracy percentages reflect better cognitive control, attentional capacity, and inhibitory function.
  Performance in the incongruent condition is of particular interest, as it requires greater cognitive effort and executive control.
Cognitive Function: N-Back | Baseline (Week 0),Week 1 (after 3 sessions), Week 6 (post-intervention, after session 18)
  The N-Back Test is a cognitive task designed to assess working memory, attention, and cognitive flexibility. It requires participants to continuously monitor a sequence of stimuli (e.g., letters, numbers, or shapes) and determine whether the current stimulus matches one presented N steps earlier in the sequence. The task increases in difficulty as N increases, demanding greater mental effort to update and maintain information in working memory.
  -Score Range: Accuracy Percentage (%): Proportion of correct responses over total trials. Reaction Time (ms): Time taken to respond to correct matches.
  -Interpretation: Higher accuracy reflects better working memory capacity and attentional control.
  Faster reaction times indicate efficient cognitive processing. Performance decline in higher N levels suggests increased cognitive load and reduced working memory capacity.
  Deficits in accuracy or reaction time may indicate difficulties in executive function and attentional flexibility.
Cognitive Function:Operation Span Test Task | Baseline (Week 0),Week 1 (after 3 sessions), Week 6 (post-intervention, after session 18)
  The Operation Span (O-Span) Test is a cognitive task designed to assess working memory capacity and attentional control. It requires participants to simultaneously process and store information, challenging their ability to maintain and manipulate information while handling a secondary task.
  The test includes:
  Two training trials for familiarization. Six experimental trials, with letter sequences ranging from four to six letters.
  -Score Range: Absolute Span Score: 0 to 12 (number of correctly recalled letter sequences).
  Interpretation:
  Higher scores indicate greater working memory capacity and better attentional control.
  Lower scores may suggest difficulties in managing cognitive load and maintaining task-relevant information under distraction.
  Performance reflects the ability to simultaneously process and store information, which is critical for complex cognitive tasks such as reasoning, problem-solving, and multitasking.
Cognitive Function: The Trail Making Test | Baseline (Week 0), Week 1 (after 3 sessions), Week 6 (post-intervention, after session 18)
  The Trail Making Test (TMT) is a widely used neuropsychological assessment designed to evaluate processing speed, cognitive flexibility, attention, and executive functioning.
  It consists of two parts:
  * TMT-A: Measures visual scanning, processing speed, and motor function. Participants connect numbers in ascending order (e.g., 1 → 2 → 3) as quickly as possible.
  * TMT-B: Assesses cognitive flexibility and task-switching ability. Participants alternate between numbers and letters in sequential order (e.g., 1 → A → 2 → B → 3 → C).
    * Score Range:
  Outcome Measure: Time (in seconds) taken to complete each part. Higher scores (longer times) indicate slower processing speed and reduced cognitive flexibility.
  -Interpretation: Lower scores (faster completion time) indicate better processing speed, visual attention, and cognitive flexibility.
  Higher scores (longer completion time) may reflect impairments in executive function, attention, or visuomotor speed.
Cerebral Oxygenation - Oxyhemoglobin (O₂Hb) | Baseline (Week 0), Week 1 (after 3 sessions), Week 6 (post-intervention, after session 18)
  * Method: Near-Infrared Spectroscopy (NIRS)
  * Measure: Oxyhemoglobin (O₂Hb), expressed in micromolar concentration (µM)
  * Interpretation: Higher O₂Hb levels indicate greater oxygen availability and delivery to brain tissues.
Cerebral Oxygenation - Deoxyhemoglobin (HHb) | Baseline (Week 0), Week 1 (after 3 sessions), Week 6 (post-intervention, after session 18)
  * Method: Near-Infrared Spectroscopy (NIRS)
  * Measure: Deoxyhemoglobin (HHb), expressed in micromolar concentration (µM)
  * Interpretation: Elevated HHb levels may suggest reduced oxygen extraction or utilization, potentially indicating impaired cerebral oxygenation.
Cerebral Oxygenation - Total Hemoglobin (tHb) | Baseline (Week 0), Week 1 (after 3 sessions), Week 6 (post-intervention, after session 18)
  * Method: Near-Infrared Spectroscopy (NIRS)
  * Measure: Total Hemoglobin (tHb), expressed in micromolar concentration (µM)
  * Interpretation: Higher tHb values reflect greater blood volume in cerebral tissue, which may indicate increased cerebral perfusion.
Biomarker Analysis-Vascular Endothelial Growth Factor (VEGF) Levels | Baseline (Week 0), Week 1 (after 3 sessions), Week 6 (post-intervention, after session 18)
  * Method: Enzyme-Linked Immunosorbent Assay (ELISA)
  * Unit of Measure: pg/mL
  * Interpretation: Increased VEGF levels suggest enhanced angiogenesis, vascular function, and cerebral blood flow.
Biomarker Analysis -Irisin Levels | Baseline (Week 0), Week 1 (after 3 sessions), Week 6 (post-intervention, after session 18)
  * Method: Enzyme-Linked Immunosorbent Assay (ELISA)
  * Unit of Measure: ng/mL
  * Interpretation: Higher irisin levels indicate improved metabolic regulation, muscle-derived neuroprotection, and brain function.
Biomarker Analysis-Hypoxia-Inducible Factor-1 Alpha (HIF-1α) Pathway Activation | Baseline (Week 0), Week 1 (after 3 sessions), Week 6 (post-intervention, after session 18)
  * Method: Quantitative Polymerase Chain Reaction (qPCR) / Western Blot
  * Unit of Measure: Relative expression level (fold change compared to baseline)
  * Interpretation: Increased HIF-1α activation suggests enhanced cellular adaptation to hypoxia, improved metabolic regulation, and potential neuroprotection.

SECONDARY OUTCOMES:
Autonomy and Daily Functioning (Activities of Daily Living Scale) | Baseline, and post-intervention (week 6, session 18)
  * Full Name: Activities of Daily Living (ADL) Scale
  * Description: This scale assesses an individual's ability to perform essential daily activities independently. It evaluates functions such as dressing, bathing, eating, mobility, toileting, and grooming.
  * Score Range: 0 to 6
  * Interpretation: A higher score indicates greater independence, while a lower score reflects higher dependency in daily functioning.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schega L, Peter B, Brigadski T, Lessmann V, Isermann B, Hamacher D, Torpel A. Effect of intermittent normobaric hypoxia on aerobic capacity and cognitive function in older people. J Sci Med Sport. 2016 Nov;19(11):941-945. doi: 10.1016/j.jsams.2016.02.012. Epub 2016 Apr 26. PMID 27134133
- [Background] Boulares A, Pichon A, Faucher C, Bragazzi NL, Dupuy O. Effects of Intermittent Hypoxia Protocols on Cognitive Performance and Brain Health in Older Adults Across Cognitive States: A Systematic Literature Review. J Alzheimers Dis. 2024;101(1):13-30. doi: 10.3233/JAD-240711. PMID 39093075
- [Background] Schega L, Peter B, Torpel A, Mutschler H, Isermann B, Hamacher D. Effects of intermittent hypoxia on cognitive performance and quality of life in elderly adults: a pilot study. Gerontology. 2013;59(4):316-23. doi: 10.1159/000350927. Epub 2013 May 3. PMID 23652274